CLINICAL TRIAL: NCT04650334
Title: Developing a Tailored Implementation Plan for Collaborative Care of Perinatal Depression in Vietnam
Brief Title: Collaborative Care for Perinatal Depression Care in Vietnam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ian Bennett, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00007369; R21MH122345 (NIH)
Record Dates: First submitted 2020-06-16; First posted 2020-12-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Perinatal Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perinatal Collaborative Care (Other): Experimental: Perinatal Collaborative Care in Can Tho, Vietnam This is an active treatment arm consisting of 3 health centers receiving training in collaborative care and enrollment of a total of 100 perinatal patients into collaborative care.
  Interventions: Behavioral: Collaborative Care

INTERVENTIONS:
Behavioral: Collaborative Care — Health services intervention to implement a team based model of care for perinatal depression.
  Other Names: Thinking Healthy

SUMMARY:
Depression is the most common medical disorder of pregnancy, and suicide, most frequently found in women with depression, is a major source of maternal mortality. Perinatal depression affects approximately 15% of women in pregnancy and the year postpartum and affects both women and their children, both medically and as a result of impairment in the ability to care for self and others. In low- and middle-income countries (LMICs) where food insecurity can be severe, growth stunting is seen among the infants of women with untreated depression. Fortunately, effective treatment of perinatal depression with antidepressant medications and evidence-based psychosocial interventions (such as collaborative care) mitigates these risks. Yet there are a range of obstacles within LMICs to the delivery of services for perinatal depression and maternal suicide prevention, including a lack of awareness of this disorder and related evidence-based treatments, stigma among patients and providers, scarcity of specialty mental health care providers, and the lack of health information technology supports for the longitudinal care of chronic illness.

DETAILED DESCRIPTION:
The investigators plan to use a participatory approach to systematically identify and adapt key elements of evidence-based models of perinatal depression care delivery to the cultural and health services context of Can Tho, Vietnam. Over the two-year study period the investigators will first develop a model, adapted from evidence-based approaches, for screening and treatment for women receiving perinatal care in community health centers as well as obstetric hospitals. Simultaneous exploration of potential implementation strategies to support and sustain this model in context will be identified along with the creation of a training and implementation toolkit for this setting. Using these strategies and tools the investigators will then carry out a pilot perinatal collaborative care study in a public health center and the prenatal care practice of the Can Tho Obstetric and Gynecologic Hospital. The results of this pilot will be used to revise and enhance the treatment model and related implementation tools. These will be used in subsequent trials of effectiveness and/or implementation broadly in the health care system of Can Tho. The investigators propose a mixed methods and participatory action research (PAR) developmental approach to tailor the standard collaborative care approach for the Can Tho city region of southern Vietnam. A linked capacity development program will work to develop the research skills of the Can Tho University of Medicine and Pharmacy (CTUMP) team through structured activities and interactions with investigators from the University of Washington.

Specific Aims: The specific aims of this proposed work, to be carried out over 2 years in health centers delivering perinatal care, are:

Aim 1 (Phase 1, months 1-12) Develop a tailored form of the collaborative care model of perinatal depression for the Can Tho health system context and an associated implementation plan and toolkit:

1. Carry out a participatory development effort to inform a collaborative care model for depression care and suicide prevention tailored to the existing health system infrastructure;
2. Identify potential strategies to support large scale implementation of this adapted model;
3. Develop an implementation toolkit to support this implementation.

Aim 2 (Phase 2 and Phase 3, months 13-24) Carry out a prospective pilot implementation study of the tailored collaborative care model and implementation approach:

1. Implement this model in perinatal care settings to assess the acceptability, feasibility, and costs of the model implementation toolkit via process and clinical outcome measures;
2. Revise and re-assess the model and implementation toolkit.

Aim 3 (Phase 1-3, months 1-24) Develop capacity in the Can Tho investigator team related to implementation science strategies to improve mental health care delivery:

1. Provide ongoing remote training of junior faculty at the CTUMP through ongoing feedback and involvement in the research efforts, completion of remote implementation research training, a monthly publication development meeting, and a journal club;
2. Conduct an annual in-person/virtual training addressing behavioral health integration and implementation science in Can Tho, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* eligible to be screened for depression during pregnancy and 1 year post partum

Exclusion Criteria:

* Severe mental illness

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Screening rates for perinatal depression | 4 months
  The rates of screening for perinatal depression by the clinical team will be determined. The rates of reported scores on the validated Vietnamese translation of the Patient Health Questionnaire - 9 item (PHQ-9) measure will be recorded for women receiving care at the study clinics. The scale ranges from 0-27 and a higher score is worse than lower however the completion of the survey is all that is required for this measure and not the total score. Women eligible for screening are those in pregnancy and 12 months postpartum. A total of 4 screenings are expected in this period - one in the first two trimesters of pregnancy and one in the third trimester and one in each of the six month periods following delivery. The rate will be reported for all eligible women (those in each of the above periods) who received a screening.
Rates of weekly use of a patient registry for systematic case review. Adherence to weekly use of patient registry for systematic case review | 4 months
  The use of the Care Manager Tracking System patient registry for weekly systematic case reviews will be assessed. Updated cases within the registry, preparation for case review, and documentation of treatment changes of patients will be assessed. The use of this tool for each week of the pilot study will be assessed.
Patient participation in Thinking Healthy treatment | 4 months
  The number of women who screen positive for risk of perinatal depression (PHQ-9 greater than or equal to 10) who agree to participate in the Thinking Healthy treatment program.
Persistence in Thinking Healthy treatment | 4 months
  The rate of women who agree to participate in the Thinking Healthy treatment who complete all treatment sessions.

SECONDARY OUTCOMES:
Rate of clinical improvement in depression symptom scores | 4 months
  Depression symptom scores among patients will be collected using the Patient Health Questionnaire - 9 item (PHQ-9) measure. This scale allows scores from 0-27 and a higher score is worse (greater symptomatology). The rate of patients with 50% reduction in symptoms will be determined as a measure of clinically significant improvement.

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - My Khanh Commune Health Center, Can Tho
  - Tan Thoi Commune Health Center, Can Tho

IPD SHARING:
Plan to Share IPD: Undecided